CLINICAL TRIAL: NCT06120530
Title: Effect of Intraperitoneal Bupivacaine on Postoperative Pain Control in Patients Undergoing Pelvic Organ Prolapse Repair
Brief Title: Intraperitoneal Bupivacaine for Pelvic Organ Prolapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, James Ryan Stewart, Assistant Professor of Clinical Obstetrics & Gynecology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17120
Record Dates: First submitted 2023-07-29; First posted 2023-11-07 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intraperitoneal bupivacaine (Active Comparator): 30 mL of bupivacaine without epinephrine 0.25%
  Interventions: Drug: Bupivacaine
- placebo (Placebo Comparator): Saline
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Bupivacaine — Intraperitoneal Bupivicaine without epinephrine 30 mg administered following completion of pelvic organ prolapse repair.
  Arms: Intraperitoneal bupivacaine
Other: Saline — Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effects of 30 mL intraperitoneal Bupivacaine without epinephrine 0.25% on postoperative pain control in patients undergoing pelvic organ prolapse repair. The investigators hypothesize that use of intraperitoneal Bupivacaine will decrease postoperative pain scores and opiate consumption in the postoperative period, following pelvic organ prolapse repair.

ELIGIBILITY:
4.1 Inclusion Criteria

List the criteria:

* Age >= 18 years
* Access to cell phone with text messaging capabilities (for same day surgery discharge)
* Patients undergoing pelvic organ prolapse repair with peritoneal access 4.2 Exclusion Criteria

List the criteria:

* Bupivacaine allergy
* History of epilepsy or other seizure disorder
* EKG demonstrating asymptomatic sinus bradycardia <40 bpm, symptomatic sinus bradycardia <60 bpm, first degree AV block, second degree AV block, third degree AV block, prolonged QT, atrial fibrillation, supraventricular tachycardia, or myocardial infarction
* Chronic liver disease proved by any ALT or AST elevation greater than 2x upper limit of normal
* Serum bilirubin elevation in excess of 5 mg/dL
* G6PD deficiency
* Weight less than 100 lbs
* Chronic opiate use

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Stewart, Principal Investigator — Indiana University
Locations (1):
- IU north, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melnyk M, Casey RG, Black P, Koupparis AJ. Enhanced recovery after surgery (ERAS) protocols: Time to change practice? Can Urol Assoc J. 2011 Oct;5(5):342-8. doi: 10.5489/cuaj.11002. PMID 22031616
- [Background] Meyer LA, Lasala J, Iniesta MD, Nick AM, Munsell MF, Shi Q, Wang XS, Cain KE, Lu KH, Ramirez PT. Effect of an Enhanced Recovery After Surgery Program on Opioid Use and Patient-Reported Outcomes. Obstet Gynecol. 2018 Aug;132(2):281-290. doi: 10.1097/AOG.0000000000002735. PMID 29995737
- [Background] Pan C, Hale D, Heit M. Enhanced Recovery Protocol Enhances Postdischarge Recovery After Laparoscopic Sacrocolpopexy. Female Pelvic Med Reconstr Surg. 2021 Nov 1;27(11):667-671. doi: 10.1097/SPV.0000000000001042. PMID 34171879
- [Background] Mehr AA, Elmer-Lyon C, Maetzold E, Bradley CS, Kowalski JT. Effect of Enhanced Recovery Protocol on Opioid Use in Pelvic Organ Prolapse Surgery. Female Pelvic Med Reconstr Surg. 2021 Dec 1;27(12):e705-e709. doi: 10.1097/SPV.0000000000001114. PMID 34807884
- [Background] Hota LS, Warda HA, Haviland MJ, Searle FM, Hacker MR. Opioid use following gynecologic and pelvic reconstructive surgery. Int Urogynecol J. 2018 Oct;29(10):1441-1445. doi: 10.1007/s00192-017-3474-5. Epub 2017 Sep 9. PMID 28889218
- [Background] Reagan KML, Boyles SH, Brueseke TJ, Linder BJ, Willis-Gray MG, Cichowski SB, Long JB. Postoperative Opioid Prescribing After Female Pelvic Medicine and Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2021 Nov 1;27(11):643-653. doi: 10.1097/SPV.0000000000001113. PMID 34669653
- [Background] Struller F, Weinreich FJ, Horvath P, Kokkalis MK, Beckert S, Konigsrainer A, Reymond MA. Peritoneal innervation: embryology and functional anatomy. Pleura Peritoneum. 2017 Dec 1;2(4):153-161. doi: 10.1515/pp-2017-0024. PMID 30911646
- [Background] SHEAR L, SWARTZ C, SHINABERGER JA, BARRY KG. KINETICS OF PERITONEAL FLUID ABSORPTION IN ADULT MAN. N Engl J Med. 1965 Jan 21;272:123-7. doi: 10.1056/NEJM196501212720303. No abstract available. PMID 14224216
- [Background] Moiniche S, Jorgensen H, Wetterslev J, Dahl JB. Local anesthetic infiltration for postoperative pain relief after laparoscopy: a qualitative and quantitative systematic review of intraperitoneal, port-site infiltration and mesosalpinx block. Anesth Analg. 2000 Apr;90(4):899-912. doi: 10.1097/00000539-200004000-00024. PMID 10735797
- [Background] Lowenstein L, Zimmer EZ, Deutsch M, Paz Y, Yaniv D, Jakobi P. Preoperative analgesia with local lidocaine infiltration for abdominal hysterectomy pain management. Eur J Obstet Gynecol Reprod Biol. 2008 Feb;136(2):239-42. doi: 10.1016/j.ejogrb.2006.11.008. Epub 2006 Dec 18. PMID 17178187
- [Background] Zacharakis D, Prodromidou A, Douligeris A, Athanasiou S, Hadzilia S, Kathopoulis N, Athanasiou V, Grigoriadis T. Preemptive Infiltration of Local Anesthetics During Vaginal Hysterectomy: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Urogynecology (Phila). 2022 Oct 1;28(10):667-678. doi: 10.1097/SPV.0000000000001221. Epub 2022 Jun 27. PMID 35759786
- [Background] Zahiri Sorouri Z, Milani F, Heidarzadeh A, Akhavan Azari M. Intraperitoneal Instillation of Lidocaine for Postoperative Pain Relief after Total Abdominal Hysterectomy: A Double Blinded Randomized Placebo-controlled Trial. Iran J Pharm Res. 2020 Spring;19(2):317-322. doi: 10.22037/ijpr.2020.1101084. PMID 33224238
- [Background] Visalyaputra S, Lertakyamanee J, Pethpaisit N, Somprakit P, Parakkamodom S, Suwanapeum P. Intraperitoneal lidocaine decreases intraoperative pain during postpartum tubal ligation. Anesth Analg. 1999 May;88(5):1077-80. doi: 10.1097/00000539-199905000-00020. PMID 10320172
- [Background] Safari S, Rokhtabnak F, Djalali Motlagh S, Ghanbari Garkani M, Pournajafian A. Effect of intraperitoneal bupivacaine on postoperative pain in laparoscopic bariatric surgeries. Surg Obes Relat Dis. 2020 Feb;16(2):299-305. doi: 10.1016/j.soard.2019.10.028. Epub 2019 Nov 7. PMID 31836291
- [Background] Elhakim M, Elkott M, Ali NM, Tahoun HM. Intraperitoneal lidocaine for postoperative pain after laparoscopy. Acta Anaesthesiol Scand. 2000 Mar;44(3):280-4. doi: 10.1034/j.1399-6576.2000.440310.x. PMID 10714840
- [Background] Williams DJ, Walker JD. A nomogram for calculating the maximum dose of local anaesthetic. Anaesthesia. 2014 Aug;69(8):847-53. doi: 10.1111/anae.12679. Epub 2014 May 12. PMID 24820093
- [Background] Kahokehr A, Sammour T, Vather R, Taylor M, Stapelberg F, Hill AG. Systemic levels of local anaesthetic after intra-peritoneal application--a systematic review. Anaesth Intensive Care. 2010 Jul;38(4):623-38. doi: 10.1177/0310057X1003800404. PMID 20715724
- [Background] Bahrami, Z H, et al. "Evaluation of Lidocaine and Bupivacaine in Post Operation Pain after Abdominal Hysterectomy." Journal of Mazandaran University of Medical Sciences, vol. 16, no. 53, Aug. 2006, pp. 1-8., http://jmums.mazums.ac.ir/article-1-899-en.html.
- [Background] Shalan, Hesham, et al. "Effect of Intraperitoneal Bupivacaine on Postoperative Pain Following Laparoscopic Pelvic Surgery." Gynaecological Endoscopy, vol. 11, no. 6, 2002, pp. 371-375., https://doi.org/10.1111/j.1365-2508.2002.00557.x.
- [Background] Datta, Pramatha Nath, and Arijit Roy. "Role of Intraperitoneal Instillation of Bupivacaine after Laparoscopic Cholecystectomy for Post-Operative Pain Management: A Randomized Controlled Trial." International Surgery Journal, vol. 7, no. 10, 2020, p. 3239., https://doi.org/10.18203/2349-2902.isj20203986.
- [Background] Al Kizwini, Ghassan. "Intra-Peritoneal Xylocaine Spraying for Postoperative Pain Control in Laparoscopic Cholecystectomy: A Prospective Study at Al-Yarmouk Teaching Hospital." Mustansiriya Medical Journal, vol. 16, no. 3, Dec. 2017, pp. 83-90., https://www.iasj.net/iasj/download/85fb88f576d0dfbc.
- [Background] Alemrajabi, Mahdi, et al. "Intraperitoneal Lavage with Bupivacaine 0.2% and Post-Operative Pain in Laparoscopic Colorectal Surgery: A Prospective, Double-Blind, Randomized Controlled Trial." Journal of Kerman University of Medical Sciences, vol. 27, no. 6, 29 Sept. 2020, pp. 510-519., https://doi.org/10.22062/JKMU.2020.91526.
- [Background] Darwish, Atef M., and Zein E. Zareh Hassan. "Intraperitoneal Bupivacaine vs. Tramadol for Pain Relief Following Day Case Laparoscopic Surgery." Gynaecological Endoscopy, vol. 8, no. 3, 1999, pp. 169-173., https://doi.org/10.1046/j.1365-2508.1999.00249.x.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants underwent pelvic organ prolapse surgery at one academic medical center from August 16, 2023, to March 14, 2024.
Groups:
- Intraperitoneal Bupivacaine: This arm received 30 mL of 0.25% bupivacaine without epinephrine via intraperitoneal lavage throughout the pelvis immediately prior to loss of peritoneal access.
- Placebo: This arm received 30 mL of placebo (saline) via intraperitoneal lavage throughout the pelvis immediately prior to loss of peritoneal access.
Period: Overall Study
Arm/Group | Intraperitoneal Bupivacaine | Placebo
Started | 44 | 47
Completed | 44 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraperitoneal Bupivacaine | Placebo | Total
Number analyzed (Participants) | 44 | 47 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (12.3) | 57.9 (11.7) | 57.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 47 | 91
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 43 | 46 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 44 | 44 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (4.68) | 28.7 (4.25) | 28.9 (4.47)
Smoking status [Count of Participants; unit: Participants]
  Current | 5 | 6 | 11
  Former | 11 | 8 | 19
  Never | 28 | 33 | 61
Menopausal status [Count of Participants; unit: Participants]
  Postmenopausal | 28 | 30 | 58
  Premenopausal | 16 | 17 | 33
Primary surgical intervention [Count of Participants; unit: Participants]
  Uterosacral ligament suspension | 14 | 16 | 30
  Sacrocolpopexy | 30 | 31 | 61
Concomitant surgeries [Count of Participants; unit: Participants]
  Vaginal hysterectomy | 15 | 15 | 30
  Laparoscopic hysterectomy | 5 | 8 | 13
  Robotic assisted laparoscopic hysterectomy | 13 | 11 | 24
  Salpingectomy | 15 | 18 | 33
  Salpingo-oophorectomy | 17 | 18 | 35
  Midurethral sling | 25 | 34 | 59
  Urethral bulking | 3 | 0 | 3
  Anterior colporrhaphy | 10 | 9 | 19
  Posterior colporrhaphy | 30 | 34 | 64
  Posterior vaginal mesh placement | 9 | 11 | 20
  Enterocele repair | 29 | 33 | 62
  Cystoscopy | 44 | 47 | 91
  Suprapubic catheter | 15 | 18 | 33
  Other | 6 | 5 | 11
Stage of prolapse [Count of Participants; unit: Participants] — Pelvic organ prolapse is staged from 0-4 based on the maximal extent of the prolapse leading edge. Stage 0 is no prolapse. Stage 1 is defined as the most distal part of the prolapsed organ is more than 1 cm above the hymen. Stage 2 is defined as the most distal part of the prolapsed organ is between 1 cm above and 1 cm below the hymen. Stage 3 is defined as the most distal part of the prolapsed organ is more than 1 cm below the hymen, but not within 2 cm of the total vaginal length. Stage IV is defined as the most distal part of the prolapse being within 2 cm of the total vaginal length.
  Participants
    Stage 1 | 1 | 1 | 2
    Stage 2 | 19 | 19 | 38
    Stage 3 | 23 | 21 | 44
    Stage 4 | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 4 Hours
Description: Patient pain will be measured by means of a numeric rating scale (scale from 0-10 with lower numbers indicating less pain and higher numbers indicating more pain) at 4 hours after surgical pelvic organ prolapse repair
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intraperitoneal Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 47
score on a scale | 3.16 (2.68) | 3.77 (2.52)

2. Secondary Outcome: Pain Score at 8 Hours, 12 Hours and 24 Hours
Description: Pain scores as determined by numeric rating scale (scale from 0-10 with lower numbers indicating less pain and higher numbers indicating more pain) at approximately 8, 12 and 24 hours
Time Frame: 8 hours, 12 hours and 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intraperitoneal Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 47
score on a scale
  8-hour | 3.27 (3.04) | 3.30 (2.37)
  12-hour | 2.84 (2.59) | 2.96 (1.94)
  24-hour | 3.00 (2.41) | 2.37 (1.98)

3. Secondary Outcome: Total Opiate Consumption
Description: Total opiate consumption postoperatively while inpatient as determined by morphine milligram equivalents (MME)
Time Frame: First 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents
Arm/Group | Intraperitoneal Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 47
Morphine milligram equivalents | 25.4 (22.4) | 22.0 (16.4)

4. Secondary Outcome: Time to First Narcotic
Description: Time to first narcotic dose during inpatient stay
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Intraperitoneal Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 47
Minutes | 98.0 (38.6) | 96.0 (28.3)

5. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intraperitoneal Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 47
Days | 1.0 (0) | 1.0 (0.15)

ADVERSE EVENTS:
Time Frame: up to 6 weeks after surgery
Arm/Group | Intraperitoneal Bupivacaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/47
Other Adverse Events (participants affected / at risk) | 4/44 | 1/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraperitoneal Bupivacaine (N=44) | Placebo (N=47)
Other (Renal and urinary disorders) | 1 | 1 — Postoperative incomplete bladder emptying
Other (Renal and urinary disorders) | 1 | 0 — Postoperative acute kidney injury suspected to be from hypovolemia during surgery.
Other (Gastrointestinal disorders) | 1 | 0 — Postoperative ileus
Other (Skin and subcutaneous tissue disorders) | 1 | 0 — Rash suspected to be from surgical drapes

LIMITATIONS AND CAVEATS:
Limitations of this study include the lack of preoperative baseline pain assessment. Additionally, because pain assessments were obtained based on surgery end time, there is likely some variability in the time interval between intervention administration and pain assessment. Lastly, time to first narcotic dose could only be assessed among those that required opioids inpatient, thus resulting in lower power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT06120530/Prot_SAP_000.pdf